CLINICAL TRIAL: NCT06951971
Title: A Multiple Center, Prospective, Single Arm, Phase III Clinical Study to Evaluate the Efficacy and Safety of Dose-modified Emapalumab and Ruxolitinib in the Treatment of Hemophagocytic Lymphohistiocytosis
Brief Title: Dose-modified Emapalumab and Ruxolitinib (E-Ru) Regimens for Hemophagocytic Lymphohistiocytosis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Xuefeng He, The First Affiliated Hospital of Soochow University, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-Ru
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hemophagocytic Lymphohistiocytosis (HLH)
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Salvage Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-Ru for HLH (Experimental): dose-modified Emapalumab+Ruxolitinib for the treatment of HLH patients.
  Interventions: Drug: dose-modified E-Ru; Other: Salvage treatment and follow-up

INTERVENTIONS:
Drug: dose-modified E-Ru — Emapalumab (1-2 mg/kg intravenously once weekly for 8 weeks) + Ruxolitinib (15-30 mg orally twice daily for 8 weeks)
Other: Salvage treatment and follow-up — 1) for patients who did not respond to the E-Ru regimen after 7 days or who relapsed at any point during treatment, a rescue regimen such as HLH-94 or doxorubicin-etoposide-methylprednisolone (DEP) was administered; 2) for patients diagnosed with lymphoma after enrollment, chemotherapy was initiated; 3) for patients who completed 8 weeks of treatment without recurrence and had no detected HLH-related gene mutations, follow-up was initiated; and 4) for patients who met the criteria for allo-HSCT, allo-HSCT was performed.

SUMMARY:
This study is trying to evaluate the efficacy and safety of dose-modified Emapalumab and Ruxolitinib (E-Ru) regimens for the treatment of active hemophagocytic lymphohistiocytosis.

DETAILED DESCRIPTION:
This clinical trial is designed to evaluate a new treatment strategy for patients with active Hemophagocytic Lymphohistiocytosis (HLH)-a rare but severe immune disorder characterized by excessive inflammation and immune system activation. HLH can be life-threatening if not treated effectively.

The study is prospective and multicenter, meaning it will be conducted at multiple hospitals and medical institutions, and patients will be followed over time to assess treatment outcomes.

We aim to test the combination of two medications:

1. Emapalumab, a monoclonal antibody that blocks interferon-gamma, a key driver of the overactive immune response seen in HLH. In this trial, it will be used at a lower-than-standard dose to reduce potential side effects.
2. Ruxolitinib, a JAK1/2 inhibitor that can reduce inflammation by interfering with immune signaling pathways. It will be administered at a higher-than-standard dose to enhance its therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfillment of at least five of the eight HLH-2004 criteria for HLH;
2. Age 1-70 years old;
3. No prior chemotherapy for HLH;
4. Confirmed not pregnant and willing to use effective contraceptive measures during the study period, with the last dose of medication administered at least 12 months prior;
5. Signed informed consent prior to study participation.

Exclusion Criteria:

1. According to the New York Heart Association (NYHA) score, patients with heart disease of grade II or above (including grade II);
2. HIV-infected patients;
3. Patients with severe renal dysfunction (glomerular filtration rate <15 mL/min);
4. Patients with severe liver cirrhosis (MELD score>20);
5. Uncontrollable infections (including lung infections, intestinal infections, etc.);
6. Have serious mental illness;
7. Have a history of active tumor;
8. Participate in other clinical investigators at the same time;
9. People with central nervous system involvement;
10. Exclusion criteria related to concomitant medication.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
60-days OS | 60 days
  overall survival (OS) rate at 60 days (2-month OS)

SECONDARY OUTCOMES:
Response rate | 7, 14, 28, and 56 days
  The ORR was defined as the percentage of patients with a complete response (CR), a partial response (PR), or an improvement in the measures of HLH.
Security | 7, 14, 28, and 56 days
  Adverse events (AEs) were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE 5.0).
EFS | 6 months
  event-free survival, defined as the time from the first administration of E-Ru until no response on day 7, disease progression or death from any cause
Overall survival | 6 months
  OS (defined as the time from the first administration of E-Ru until death from any cause)
Trend of related indicators | 7, 14, 28, and 56 days
  Changes in biomarkers between baseline and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng He, Dr., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided